CLINICAL TRIAL: NCT06627634
Title: Gastric Cancer and Oligometastatic Liverinvolvement. Metastatectomy and Impact on Survival
Brief Title: Radical Surgery for Advanced Gastric- or GEJ-cancer With Oligometastatic Dissmination to the Liver
Acronym: LEVECA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Julie Lykke Harbjerg, MD, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-233-20
Record Dates: First submitted 2023-05-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients with oligometastatic spread form gastric og GEJ-cancer are offered standart curative treatment along with metastatectomia in the liver.
  Interventions: Procedure: Metastatectomia and standard treatment for resectable disease.

INTERVENTIONS:
Procedure: Metastatectomia and standard treatment for resectable disease. — Rather than palliative chemotherapy, the intervention offered to participants is preoperative chemotherapy, resection of primary tumour and metastatectomia of oligometastatic spread to the liver. If fit for post-operative chemotherapy, this is offered as well.

SUMMARY:
Offering treatment with potential to cure for participants with no such offer in today's standard treatment options, by offering metastatectomia and standard treatment with intention to cure i.e., neoadjuvant chemotherapy and gastrectomy for participants with gastric- og gastroeusofageal junction cancer. Including 20 participants from all 4 centres in Denmark able to perform the surgical procedures in question.

Endpoints: 2-year overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18.
* Presence of primary T1-T4N0-N3M1 adenocarcinoma of the stomach or GEJ and max. 30% liver involvement.
* Primary tumour resectable, based on imaging workup.
* Surgical operable patients with ASA-score36 ≤ III and WHO performance status37 0-1.
* Patients eligible for treatment with systemic chemotherapy by FLOT regimen.
* Informed consent is obtained.

Exclusion Criteria:

* Patient with non-resectable cancer.
* Direct growth involving adjacent organs, i.e., pancreas, colon, blood vessels or bones.
* Other malignant disease diagnosed or treated up to 2 years prior to inclusion, except non-aggressive cancers such as non-melanoma sin cancer.
* Altered anatomy of the upper gastrointestinal tract due to previous surgery of the oesophagus, stomach, and duodenum.
* BMI ≤ 18
* The patient is unable to understand and/or read the consent form.
* Other serious illness or acute infections.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Willy Kjaer, MD, PhD, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus Univercity hospital, Aarhus, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No